CLINICAL TRIAL: NCT03598959
Title: Phase I/II Study of Safety and Efficacy of Tofacitinib Combined With Chidamide in Patients With Relapsed and Refractory Extranodal Natural Killer/T Cell Lymphoma
Brief Title: Tofacitinib Combined With Chidamide in R/R ENKTCL
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sichuan University (Other)
Responsible Party: Principal Investigator, Jie Ji, Clinical Professor, Sichuan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HXNKT 2.0
Record Dates: First submitted 2018-07-16; First posted 2018-07-26 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Extranodal NK/T-cell Lymphoma
MeSH Terms: conditions — Lymphoma, Extranodal NK-T-Cell | interventions — tofacitinib; N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (Experimental): Treated with tofacitinib and chidamide for 4 cycles.
  Interventions: Drug: tofacitinib; Drug: chidamide

INTERVENTIONS:
Drug: tofacitinib — orally 10 mg daily
Drug: chidamide — orally 20 mg twice weekly

SUMMARY:
This study is to explore the efficacy and safety of tofacitinib combined with chidamide in patients with relapsed and refractory extranodal NK/T cell lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients with primary refractory or recurrent extranodal NK/T cell lymphoma that do not qualify for treatment protocols of higher priority.

  2. Adequate renal function, as defined by estimated serum creatinine clearance >/=50 ml/min and/or serum creatinine </= 1.8 mg/dL.

  3. Adequate hepatic function, as defined by serum glutamate oxaloacetate transaminase (SGOT) and/or serum glutamate pyruvate transaminase (SGPT) </= 3 x upper limit of normal; serum bilirubin and alkaline phosphatase </= 2 x upper limit of normal.

  4.. Adequate cardiac function with left ventricular ejection fraction >/= 50%. No uncontrolled arrhythmias or symptomatic cardiac disease.

  5. Performance status 0-1. 6. Negative Beta diffusing capacity of lung for carbon monoxide (HCG) text in a woman with child-bearing potential, defined as not post-menopausal for 12 months or no previous surgical sterilization

Exclusion Criteria:

-1. Patients relapsed after allogeneic stem cell transplant 2. Patients with active hepatitis B or C(HBV DNA >/=10,000 copies/mL). 3. Active infection requiring parenteral antibiotics 4. HIV infection, unless the patient is receiving effective antiretroviral therapy with undetectable viral load and normal cluster of differentiation 4 (CD4) counts 5. Evidence of either cirrhosis or stage 3-4 liver fibrosis in patients with chronic hepatitis C or positive hepatitis C serology.

6. Patients with a cQT longer than 500 ms

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-01-01 (Estimated); Primary Completion 2019-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
2-year progression free survival | 2 years after recruitment

SECONDARY OUTCOMES:
complete remission | 4 months after treatment
adverse events (AEs) | 2 years after recruitment
2-year overall survival | 2 years after recruitment

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital of Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lee S, Park HY, Kang SY, Kim SJ, Hwang J, Lee S, Kwak SH, Park KS, Yoo HY, Kim WS, Kim JI, Ko YH. Genetic alterations of JAK/STAT cascade and histone modification in extranodal NK/T-cell lymphoma nasal type. Oncotarget. 2015 Jul 10;6(19):17764-76. doi: 10.18632/oncotarget.3776. PMID 25980440